CLINICAL TRIAL: NCT01217970
Title: Phase I Safety Interaction Trial of Ibudilast With Methamphetamine
Brief Title: Safety Interaction Trial Ibudilast and Methamphetamine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); MediciNova (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: ShoptawPI_ibudilast; R01DA029804 (NIH)
Record Dates: First submitted 2010-10-06; First posted 2010-10-08 (Estimated); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Methamphetamine-dependence; Substance Abuse
Keywords: methamphetamine; dependence; stimulant; amphetamine; los angeles; meth; speed; crank; abuse
MeSH Terms: conditions — Substance-Related Disorders | interventions — ibudilast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo, Ibudilast 20 mg, then Ibudilast 50mg (Experimental): Sequence: (1) Placebo, (2) Ibudilast 20 mg BID, then (3) Ibudilast 50 mg BID
  Interventions: Drug: Ibudilast 20mg; Drug: Ibudilast 50mg; Drug: Placebo oral tablet
- Ibudilast 20 mg, Ibudilast 50mg, then placebo (Experimental): Sequence: (1) Ibudilast 20 mg BID, (2) Ibudilast 50 mg BID, then (3) Placebo
  Interventions: Drug: Ibudilast 20mg; Drug: Ibudilast 50mg; Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Ibudilast 20mg — Ibudilast 20mg BID
  Other Names: IBUD
Drug: Ibudilast 50mg — Ibudilast 50mg BID
  Other Names: IBUD
Drug: Placebo oral tablet
  Other Names: Placebo

SUMMARY:
This study is designed to collect data to determine whether a medication, ibudilast, is safe for use as a potential treatment for methamphetamine-dependent people. For 18 years in Japan and South Korea, ibudilast has been used safely in humans as a treatment for asthma, pulmonary, and cardiovascular disease. It is not known whether ibudilast is safe to use in outpatient settings with people who have methamphetamine dependence. This would be the first study to collect this information. This study is important because individuals with methamphetamine dependence often relapse to meth use, even when in treatment; some number of individuals who participate in an outpatient study will relapse to methamphetamine while taking ibudilast. It is crucial to know whether there may be interactions between ibudilast and methamphetamine before planning an outpatient clinical trial.Ibudilast is an exciting medication candidate for treating methamphetamine dependence. When individuals become abstinent from methamphetamine during early recovery, the body starts an inflammatory process in neurons, especially glial cells. Glial cells are important in that they provide support to the nerve cells that are involved in thought, movement, and other human activities. By dampening inflammation in glial cells, ibudilast may preserve glial and other nerve cells during early abstinence, which in turn may help individuals feel better and think better during treatment.

The study specific aims are to determine whether ibudilast alters:

1. blood pressure and heart rate responses to methamphetamine;
2. the ratings of craving or other drug experiences from methamphetamine;
3. the reward/reinforcing effects of methamphetamine; and
4. the metabolism of methamphetamine.

Over an enrollment period of 24 months, 12 methamphetamine-dependent participants who are not looking for treatment will complete this study.

DETAILED DESCRIPTION:
This study is designed to collect data to determine whether a medication, ibudilast, is safe for use as a potential treatment for methamphetamine-dependent people. For 18 years in Japan and South Korea, ibudilast has been used safely in humans as a treatment for asthma, pulmonary, and cardiovascular disease. It is not known whether ibudilast is safe to use in outpatient settings with people who have methamphetamine dependence. This would be the first study to collect this information. This study is important because individuals with methamphetamine dependence often relapse to meth use, even when in treatment; some number of individuals who participate in an outpatient study will relapse to methamphetamine while taking ibudilast. It is crucial to know whether there may be interactions between ibudilast and methamphetamine before planning an outpatient clinical trial.

The study will be conducted at the Harbor-UCLA hospital to ensure the medical safety of participants, especially if there are unexpected interactions between ibudilast and methamphetamine on cardiovascular function. Methamphetamine can cause substantial increases in heart rate and blood pressure that last for about 3 hours. This study will measure whether people who are meth-dependent (and not looking for treatment) show increases in their heart rate and blood pressures when given methamphetamine above what is expected by methamphetamine alone and when at the recommended doses of ibudilast.

Ibudilast is an exciting medication candidate for treating methamphetamine dependence. When individuals become abstinent from methamphetamine during early recovery, the body starts an inflammatory process in neurons, especially glial cells. Glial cells are important in that they provide support to the nerve cells that are involved in thought, movement, and other human activities. By dampening inflammation in glial cells, ibudilast may preserve glial and other nerve cells during early abstinence, which in turn may help individuals feel better and think better during treatment.

The study specific aims are to determine whether ibudilast alters:

1. blood pressure and heart rate responses to methamphetamine;
2. the ratings of craving or other drug experiences from methamphetamine;
3. the reward/reinforcing effects of methamphetamine; and
4. the metabolism of methamphetamine.

Over an enrollment period of 24 months, 12 methamphetamine-dependent participants who are not looking for treatment will complete this study. Each participant will complete assessments of safety/tolerability, perceived effects of methamphetamine, and an assessment where subjects make choices between different amounts of money and methamphetamine. Each patient will stay in the hospital for a total of 27 nights. The first two days consist of safety infusions to make sure methamphetamine is tolerable. Then, each subject will start study medication and take a 7-day course of three conditions: placebo, ibudilast 20mg BID, and ibudilast 50mg ibudilast. Low dose ibudilast always precedes high dose ibudilast. The order of placebo being first or last is random.

ELIGIBILITY:
Inclusion Criteria:

1. NOT seeking treatment for methamphetamine problems;
2. English-speaking;
3. Age 18-55;
4. Meet SCID criteria for MA dependence;
5. Self-reported history of MA use via injection or smoking AND at least one MA positive urine drug screening during eligibility;
6. Resting heart rate 50-100BPM; Systolic BP 105-150 mm Hg; Diastolic BP 45-90 mm Hg stabilized within 2 days of admission;
7. Baseline EKG demonstrating normal sinus rhythm, normal conduction, no clinically significant arrhythmias;
8. Use of acceptable barrier method of birth control;
9. If female, not pregnant or lactating;
10. Have medical history and physical examination demonstrating no additional clinically significant contraindications for study participation, in judgment of investigators.

Exclusion Criteria:

1. Current dependence on cocaine, opioids, marijuana, or alcohol;
2. Liver function tests GE 3x upper limit of normal, or kidney function tests GE 2x the upper limit of normal;
3. Current or past history of seizure disorder;
4. History of head trauma;

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2011-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 35 days
  Insomnia, Nicotine craving, Gastrointestinal upset, Headache, Musculoskeletal pain, Pain at IV site, Rash, Vivid dreams, Constipation, Dizziness, Dysuria, Ectopic heart beats, Fever/chills/hot flashes, Pruritis, Sore throat, Tinnitus, Backache, Chest congestion, Sedation, or other reported by patient or observed by clinician
Number of Participants with Clinically Significant Changes in Cardiovascular Parameters as a Measure of Safety and Tolerability | 35 days
  Systolic and diastolic blood pressure, heart rate, and an EKG "rhythm strip"

SECONDARY OUTCOMES:
Number of participants with adverse outcomes on (1) VAS, drug-effect scale, subjective effects, etc., and (2) pharmacokinetics of methamphetamine as measures of efficacy | 35 days
  1. Barratt Impulsiveness Scale-11; The Wechsler Test of Adult Reading; Wender Utah Rating Scale; subjective intensity of 12 drug effects on VAS.
  2. blood concentrations of methamphetamine and amphetamine
  3. cytokine panel from plasma

CONTACTS AND LOCATIONS:
Overall Officials: Steven Shoptaw, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Harbor-UCLA Medical Center GCRC, Torrance, California, United States